CLINICAL TRIAL: NCT04027387
Title: A Phase Placebo-Controlled, Sequential Single Dose Escalation Study of the Safety, Pharmacokinetics, and Antiretroviral Activity of IVTMB-365 in HIV-1 Infected Participants
Brief Title: Dose Escalation Safety Study of TMB-365 in HIV-1 Infected Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: TaiMed Biologics Inc. (Industry)
Collaborators: Westat (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TMB-365-101
Record Dates: First submitted 2019-07-17; First posted 2019-07-22 (Actual); Last update posted 2021-10-06 (Actual); Status verified 2021-10

CONDITIONS: HIV-1-infection

STUDY DESIGN:
Intervention Model Description: Single dose escalation
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind placebo controlled. Study pharmacist unblinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- TMB-365 400 mg- Group 1 (Experimental): Single dose of TMB-365 400 mg or matching placebo by intravenous infusion
  Interventions: Biological: TMB-365
- TMB-365 800 mg- Group 2 (Experimental): Single dose of TMB-365 800 mg or matching placebo by intravenous infusion
  Interventions: Biological: TMB-365
- TMB-365 1600 mg- Group 3 (Experimental): Single dose of TMB-365 1600 mg or matching placebo by intravenous infusion
  Interventions: Biological: TMB-365

INTERVENTIONS:
Biological: TMB-365 — An IgG1 monoclonal antibody targeting domain 2 of the CD4 receptor for treatment of HIV-1 infection

SUMMARY:
This study will evaluate the safety and behavior in the body of the experimental drug TMB-365 in people with HIV-1 infection. This will be the first test of TMB-365 in humans. One dose of the study drug is given to each participant, followed by 10 weeks of monitoring for safety and levels of the drug in the blood. The first group of participants will receive the lowest dose (400 mg). If no safety concerns are seen, the next group will begin at a higher dose (800 mg). If no safety concerns are seen in the second group, the third group will begin at the highest dose in this study (1600 mg).

DETAILED DESCRIPTION:
This phase 1, randomized, double-blinded, placebo-controlled, sequential single dose escalation study will evaluate the safety, tolerability and pharmacokinetic (PK) parameters of TMB-365 administered via intravenous infusion (IV) to HIV-1 infected participants at one of three successively increasing dose levels: 400 mg, 800 mg, and 1600 mg. Each participant will be monitored for 10 weeks post-administration. All participants will be expected to participate in PK sampling during Weeks 1, 4, 5, and 6.

Beginning with the lowest dosage group, a Data Monitoring Committee (DMC) will review available data after four participants have completed two weeks of post-dose follow-up to determine if dosing of the next dosage group may proceed.

If no dose limiting toxicities (DLTs) emerge, defined as a single Grade 4 or two of the same Grade 3 clinical or laboratory adverse events deemed possibly, probably or definitely related to the study drug, or a serious adverse event deemed possibly, probably or definitely related to the study drug as graded by the DAIDS Table for Grading Severity of Adult and Pediatric Adverse Events Version 2.1, then dosing of the next higher dose group will be permitted.

Dosing in the highest dose group will begin after four of the eight participants in second group have successfully completed the scheduled study drug administration and two weeks of follow-up, and those data, along with all available data from the initial dose group have been reviewed by the DMC and no DLTs or SAEs as defined above are identified.

All participants may initiate standard combination antiretroviral therapy six weeks after receiving the study drug.

ELIGIBILITY:
Inclusion Criteria:

* Male or female at least 18 years of age and no greater than 60 years on the day of Screening
* Asymptomatic HIV-1 infection, documented by any licensed rapid HIV test or HIV enzyme or chemiluminescence immunoassay (E/CIA) test kit at any time prior to study entry and confirmed by Geenius™ or a second antibody test by a method other than the initial rapid HIV and/or E/CIA test, or by HIV-1 antigen, plasma HIV-1 RNA viral load
* Has not received ART for three months prior to the first dose.
* Screening HIV-1 RNA ≥ 1,000 copies/mL and < 100,000 copies/mL obtained within 60 days prior to the first dose.
* Laboratory values obtained within 60 days prior to the first dose:

  * Hemoglobin > 10.0 g/dL
  * Platelet count ≥ 100,000/mm3
  * Absolute neutrophil count ≥ 1,000/mm3
  * Serum aspartate aminotransferase (AST) and alanine aminotransferase (ALT) < 1.5 x upper limit of normal (ULN)
  * Creatinine clearance (CrCl) of ≥ 50 mL/min
* Willing to comply with the requirements of the protocol and available for follow-up for the planned duration of the study.
* In the opinion of the principal investigator or designee, has understood the information provided; written informed consent needs to be given before any study-related procedures are performed
* Females of childbearing potential, sexually active with a male sex partner, must agree to use one effective method of contraception from the time of signing the consent to completion of the study, and agree to pregnancy testing as per the Schedule of Events and Procedures. Females of childbearing potential are female participants who are not surgically sterile (no history of bilateral tubal ligation, hysterectomy, or bilateral salpingo-oophorectomy), are not postmenopausal (at least one year without menses), and are not otherwise sterile by medical evaluation.

Exclusion Criteria:

* Receipt of TMB-365, TROGARZO (ibalizumab-uiyk), or any anti-CD4 therapeutic (e.g., UB-421) at any time prior to the first dose
* Pregnant, planning a pregnancy during the trial period, or lactating.
* Known allergy/sensitivity or any hypersensitivity to components of the study drug or its formulation, or known allergy to a MAb
* Major psychiatric illness including any history of schizophrenia or severe psychosis, bipolar disorder requiring therapy, or suicide attempt in the previous three years
* Serious illness requiring systemic treatment and/or hospitalization within 21 days prior to the first dose
* Receipt of immunomodulatory agents (e.g., interleukins, interferons, cyclosporine, high dose systemic corticosteroids), HIV vaccine, systemic cytotoxic chemotherapy, or investigational therapy within 180 days prior to the first dose
* Any chronic or acute medical condition, including drug use and alcohol abuse, which in the opinion of the investigator would interfere with evaluation of the study drug
* Lack of adequate venous access
* Individuals who have experienced virologic failure during treatment with two or more cART treatment regimens. Note that a change in treatment regimen for intolerance is not considered treatment failure.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2019-12-14 (Actual); Primary Completion 2021-08-18 (Actual); Study Completion 2021-08-18 (Actual)

PRIMARY OUTCOMES:
Safety of a single 400mg dose of TMB-365 | 10 weeks
  % of subjects with treatment-emergent adverse events
Safety of a single 800mg dose of TMB-365 | 10 weeks
  % of subjects with treatment-emergent adverse events
Safety of a single 1600mg dose of TMB-365 | 10 weeks
  % of subjects with treatment-emergent adverse events
Pharmacokinetics of a single 400mg dose of TMB-365 | 4 weeks
  % CD4 receptor occupancy
Pharmacokinetics of a single 800mg dose of TMB-365 | 4 weeks
  % CD4 receptor occupancy
Pharmacokinetics of a single 1600mg dose of TMB-365 | 4 weeks
  % CD4 receptor occupancy

SECONDARY OUTCOMES:
Antiviral activity of a single 400 mg dose of TMB-365 | 2 weeks
  Change in log10 plasma HIV-1 RNA
Antiviral activity of a single 800 mg dose of TMB-365 | 2 weeks
  Change in log10 plasma HIV-1 RNA
Antiviral activity of a single 1600 mg dose of TMB-365 | 2 weeks
  Change in log10 plasma HIV-1 RNA

CONTACTS AND LOCATIONS:
Overall Officials: Steve Weinheimer, PhD, Study Director — TaiMed Biologics
Locations (6):
- United States (5):
  - Quest Clinical Research, San Francisco, California
  - Midway Immunology and Research Center, Ft. Pierce, Florida
  - Orlando Immunology Center, Orlando, Florida
  - University of Mississippi Medical Center Division of Infectious Diseases, Jackson, Mississippi
  - North Texas Infectious Disease Consultants, Dallas, Texas
- Clinical Research PR, Inc, San Juan, Puerto Rico

IPD SHARING:
Plan to Share IPD: No